CLINICAL TRIAL: NCT04467125
Title: Nexplanon Removal: Subcutaneous vs. Topical Lidocaine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Manish Jain, Associate Professor, Dept. of Obstetrics and Gynecology, Augusta University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1288589-4
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Contraception
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EMLA (Experimental): Subjects randomized to EMLA receive one inch of EMLA cream placed at the removal site and then have an occlusive dressing placed. One hour later they have the Nexplanon device removed.
  Interventions: Drug: Eutectic Lidocaine Prilocaine
- Subcutaneous Lidocaine (Active Comparator): Subjects randomized to subcutaneous lidocaine have 1% lidocaine injected at the removal site and then undergo Nexplanon removal.
  Interventions: Drug: Subcutaneous Lidocaine

INTERVENTIONS:
Drug: Eutectic Lidocaine Prilocaine — Subjects randomized to EMLA receive one inch of EMLA cream placed at the removal site and then have an occlusive dressing placed. One hour later they have the Nexplanon device removed.
  Other Names: EMLA
  Arms: EMLA
Drug: Subcutaneous Lidocaine — Subjects randomized to subcutaneous lidocaine have 1% lidocaine injected by the provider at the removal site in an amount decided on by the provider.
  Arms: Subcutaneous Lidocaine

SUMMARY:
A randomized trial of using EMLA cream for anesthesia to remove Nexplanon versus the standard route of subcutaneous lidocaine for anesthesia. Primary endpoints are pain during procedure and time to removal.

ELIGIBILITY:
Inclusion Criteria:

* Females with Nexplanon implant in place, desiring removal No allergy to lidocaine or any component of EMLA cream Age greater than or equal to 18years English as primary language Not pregnant

Exclusion Criteria:

* pregnant non-emglish speaking age less than 18 yo Allergy to lidocaine or EMLA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
pain of procedure | during procedure
  Using the pain scale the participant is asked to circle the numerical value of pain they had during removal.
time to perform procedure | procedure
  the medical assistant times the procedure from incision to removal of the device.

SECONDARY OUTCOMES:
How likely to recommend their anesthetic? | procedure
Provider's sense of ease of removal? | procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University Ob/Gyn Resident Continuity Clinic, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No